CLINICAL TRIAL: NCT06237894
Title: Effect of Multisensory Stimulation on Postoperative Pain, Physiological Parameters and Fear in Children After Surgical Procedure: Randomized Controlled Study
Brief Title: Multisensory Stimulation on Postoperative Pain, Physiological Parameters and Fear in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Fulya Kos, lecturer, Bilecik Seyh Edebali Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BSEU
Record Dates: First submitted 2024-01-11; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Multisensory Stimulation; Child, Only; Postoperative Pain; Fear
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multisensory Stimulation (Experimental)
  Interventions: Other: Multisensory Stimulation

INTERVENTIONS:
Other: Multisensory Stimulation — Multisensory Stimulation

SUMMARY:
It is known that non-pharmacological methods are effective in reducing pain in children and that they increase the effectiveness of drugs when used together with analgesics. Non-pharmacological methods are preferred because they are easy to apply and cheap, and they reduce the need for drug administration and thus the risk of side effects. Knowing the impact of pain and associated fear on children, developing appropriate pain control strategies is both a medical and ethical responsibility. Reviewing the literature, there is little scientific evidence that multisensory stimulation is an effective intervention in reducing pain and fear after surgery in children. When the studies on the effect of multisensory stimulation on pain and fear in childhood are examined, it is seen that the studies mostly aim to reduce pain and fear in the neonatal period or before surgery. It is thought that it is an important limitation that multisensory stimulation, which is an effective method for reducing pain and fear in childhood, does not examine its direct effects on postoperative pain, physiological parameters and fear after surgical procedures in children. In this context, the aim of the study is to examine the effect of multisensory stimulation on postoperative pain, physiological parameters and fear in children after the surgical procedure.

DETAILED DESCRIPTION:
The causes of surgery seen in childhood vary according to age. Congenital anomalies are the most common in the neonatal period, and in other age periods, the most common are gastrointestinal system (appendicitis, intussusception, inguinal hernia, etc.) and urogenital system surgeries (circumcision, hydrocele, undescended testicle, testicular torsion, hypospadias, laparoscopic interventions, ovarian cyst and torsion, etc.). They may undergo surgical procedures due to reasons such as .). In a child undergoing a surgical procedure; Postoperative complications such as apnea, airway obstruction, aspiration, extubation, laryngospasm, bronchospasm may occur. One of the most common problems seen in children after surgical procedures is pain. Studies have shown that 24-80% of children who undergo surgery are accompanied by moderate to severe pain. If postoperative pain is not relieved effectively, it may cause negative physiological effects such as increased respiration and pulse, decreased saturation, crying, restlessness, nausea and vomiting, oliguria, impaired immune response, decreased wound healing, and anorexia.

One of the most common problems seen in children after surgical procedures is fear. Postoperative pain that occurs after surgery, different environment and change of routine, different sounds, lights and equipment, unfamiliar people, painful procedures, being away from family members and friends, general anesthesia complications such as nausea and vomiting, loss of control, activity limitation. Communication difficulties, dark environments and the presence of other crying children can create fear in children. This situation can be traumatic, especially for children who have difficulty understanding what is happening to them during surgical procedures and who have difficulty coping with such situations that create fear.

In order to provide benefits such as accelerating recovery and increasing nurse-child interaction in the postoperative period, interventions such as pain management and fear reduction should be prioritized. The main purpose of pain management is; Relieving pain is minimizing the resulting fear and side effects. Opioids are the cornerstone of treatment in the field of postoperative pain management in the pediatric population. Despite the benefits and widespread use of opioids in pain management, opioids; It may cause undesirable side effects such as postoperative nausea, vomiting, urinary retention, constipation, respiratory depression, cognitive impairment, addiction, and may prolong hospital stay in children. In studies, the use of multimodal treatment is recommended due to the side effects of opioid use. A combination of pharmacological and non-pharmacological treatments has been shown to reduce dependence on opioids and their side effects, reduce acute pain symptoms and fear in the postoperative period, and increase emotional well-being. In the literature, recent studies on non-pharmacological methods to control pain and reduce fear suggest the use of multi-sensory stimulation to distract children and create a happy and motivating atmosphere.

Multi-sensory stimulation; It is a non-pharmacological method that aims to support the child's developmental stages, reduce behavioral problems, and reduce pain and fear, especially with stimulating materials for the sense of sight, hearing, smell and touch. In its basic mechanism, multisensory stimulation provides multiple stimuli by continuously activating tactile, thermal and emotional systems. This simultaneous stimulation of various sensory systems causes sensory satiation. In this way, gate-control mechanism gates are activated to weaken or suppress nociceptive transmission. Thus, the gate-control mechanism reduces or eliminates the occurrence of pain by closing the gates to prevent nociceptive messages from entering. Multi-sensory stimulation applications include; These include mother-baby communication, skin-to-skin contact, breastfeeding, which activates the sensory receptors on the skin and the sense of taste, and making the baby smell breast milk, amniotic fluid or aromatic scents that it recognizes. Establishing eye contact with the baby, speaking in a soft voice, massaging, wrapping, and using the parent's scent are among the multi-sensory stimulation practices. It is known that non-pharmacological methods are effective in reducing pain in children and that they increase the effectiveness of drugs when used together with analgesics. Non-pharmacological methods are preferred because they are easy to apply and cheap, and they reduce the need for drug administration and thus the risk of side effects. Knowing the impact of pain and associated fear on children, developing appropriate pain control strategies is both a medical and ethical responsibility. Reviewing the literature, there is little scientific evidence that multisensory stimulation is an effective intervention in reducing pain and fear after surgery in children. When the studies on the effect of multisensory stimulation on pain and fear in childhood are examined, it is seen that the studies mostly aim to reduce pain and fear in the neonatal period or before surgery. It is thought that it is an important limitation that multisensory stimulation, which is an effective method for reducing pain and fear in childhood, does not examine its direct effects on postoperative pain, physiological parameters and fear after surgical procedures in children. In this context, the aim of the study is to examine the effect of multisensory stimulation on postoperative pain, physiological parameters and fear in children after the surgical procedure.

ELIGIBILITY:
Sampling Inclusion Criteria:

* Children are between the ages of 5-10,
* Having undergone a surgical intervention,
* Does not have an additional disease/condition that will affect the child's oxygen saturation, blood pressure and heart rate,
* Two hours have passed since the last painful attempt,
* Children whose parents agree to participate in the study will be included in the study.

Exclusion Criteria from the Sample:

* Hearing and vision impaired
* Does not have a mental disability
* Children who do not have a parental consent form will not be included in the research.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Descriptive Information Form | one year
  The form prepared by the researchers in line with the literature consists of 19 questions including socio-demographic characteristics, information about the child's disease, and the parent's perception of pain and fear. This form will also record the child's physiological parameters (heart rate and oxygen saturation) during the painful procedure.
Wong Baker Faces Pain Rating Scale | one year
  This scale is rated from 0 to 10. 0 indicates no pain and 10 indicates the most severe pain. Pain is requested to be evaluated according to facial expression. The scale was developed by Donna Wong and Connie Morain Baker in 1981 and revised in 1983. This scale is used to diagnose pain in children between the ages of 3-18. Wong Baker Pain Rating Scale The guideline recommends that clinicians use a validated pain rating scale when assessing postoperative pain and adjust treatment accordingly (strong recommendation, low-quality evidence), but there is insufficient evidence on the effect of different pain rating scales on postoperative pain outcomes. Therefore, when choosing a specific pain assessment tool, factors such as developmental status, cognitive status, level of consciousness, level of education, cultural and language differences should also be taken into consideration.
Children's Fear Scale | one year
  Children's Fear Scale, the scale whose validity and reliability was established by Gerçeker et al. (2018), is used to measure the child's anxiety level. Children's Fear Scale is a scale that evaluates between 0 and 4, consisting of showing five drawn facial expressions ranging from neutral expression (0 = no fear) to scared face (4 = severe fear). Pain and anxiety before and during the procedure can be used by families and researchers to evaluate children and is intended for children between the ages of 5-10. Children's Fear Scale was created based on McKinley et al.'s (2003) Faces Anxiety Scale, which was developed to measure the fear or anxiety of adults in the intensive care unit. It is a scale consisting of one item and five gender-neutral facets. Facial muscle changes in fearful expressions were drawn by a graphic artist based on photographs of scared faces.

IPD SHARING:
Plan to Share IPD: No
No planning